CLINICAL TRIAL: NCT02370784
Title: The Effect of Atorvastatin on Microvascular Endothelial Function and Raynaud in Early Diffuse Systemic Sclerosis
Brief Title: Atorvastatin for Microvascular Endothelial Function and Raynaud in Early Diffuse Scleroderma
Acronym: TAMER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Robyn T. Domsic, MD, MPH (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor-Investigator, Robyn T. Domsic, MD, MPH, MD, MPH, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO14010170; 1R21AR066305-01A1 (NIH)
Record Dates: First submitted 2015-01-26; First posted 2015-02-25 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Scleroderma
Keywords: early diffuse scleroderma; Raynaud
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Drug (Active Comparator): atorvastatin 40 mg once daily for sixteen weeks
  Interventions: Drug: atorvastatin
- Placebo control (Placebo Comparator): receive a placebo of similar appearance once daily for sixteen weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: atorvastatin — Atorvastatin is an oral cholesterol-lowering medication commonly referred to as statin therapy.
  Other Names: Lipitor
  Arms: Active Drug
Drug: Placebo — oral drug of similar appearance to atorvastatin
  Arms: Placebo control

SUMMARY:
The purpose of this study is to learn about the effect atorvastatin on blood vessel function and Raynaud symptoms in patients with early diffuse systemic sclerosis.

Systemic sclerosis is a disease characterized by blood vessel injury, immune system activation and fibrosis. Blood vessel injury is thought to be important early in the disease. Blood vessel complications of systemic sclerosis include Raynaud phenomena, finger and toe ulcers, and pulmonary hypertension. While atorvastatin reduces cholesterol, it is recognized to have many effects beyond cholesterol reduction. These include improvement of blood vessel function and reduction of fibrosis. We hypothesize that treatment with atorvastatin over 16 weeks will improve blood vessel function and Raynaud symptom in patients with early diffuse systemic sclerosis. We hope that by targeting therapy early in the disease we may delay blood vessel changes and improve Raynaud symptoms.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a multisystem autoimmune illness characterized by vasculopathy, immune system activation and fibrosis of the skin and internal organs. SSc affects approximately 240 people per million in the US, but is a disease for which there is no FDA approved medication. Current hypothesis of pathogenesis suggest that a vascular injury with endothelial dysfunction may be an inciting event contributing to immunologic activation and fibrosis in the pathogenesis of the disease. More than 90% of individuals with SSc have vascular complications including Raynaud phenomenon, digital ulcers or gangrene and pulmonary hypertension; with microvascular abnormalities felt to contribute to Raynaud and digital ulcerations.

Statin medications are well-recognized to have pleiotropic effects which may modify all three aspects of SSc pathogenesis. Early diagnosis and treatment of microvascular endothelial dysfunction and Raynaud phenomeonan may have the greatest effect in early disease. Thus, we hypothesize that treatment with atorvastatin in a well-defined cohort of early diffuse systemic sclerosis will produce beneficial results.

Participants will be patients with early diffuse systemic sclerosis and Raynaud phenomenon who have no history of cardiovascular disease or diabetes. A total of 30 patients will be enrolled and followed for 16 weeks. Half the patients will be randomized to atorvastatin and half to placebo. Patients will be allowed to continue underlying immunosuppressive and Raynaud therapy at stable doses during the trial. Since this is a pilot study, future larger controlled trials will be necessary to clearly demonstrate drug effectiveness. Investigators are hoping that this study will give us signals to guide a future multicenter clinical trial.

ELIGIBILITY:
Inclusion Criteria:

1. early diffuse scleroderma (< 3 years from the first scleroderma-related symptom)
2. Raynaud phenomenon
3. no use of lipid-lowering medication within 60 days

Exclusion Criteria:

1. pregnancy
2. renal or kidney dysfunction (creatinine < 2.0 mg/dL or creatinine clearance < 60 c/min)
3. diabetes mellitus
4. known cardiovascular disease or a prior history of stroke
5. history of liver disease
6. new or changed dose of calcium channel blockers (CCB) and angiotensin receptor blockers (ARBs) in the last 4 weeks
7. known allergy or adverse reaction to the atorvastatin or another statin drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-02; Primary Completion 2018-12-15 (Actual); Study Completion 2019-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at a single Scleroderma Center between March 2015 and August 2017.
Groups:
- Atorvastatin 40 mg Daily: Length of intervention: 16 weeks atorvastatin: Atorvastatin is an oral cholesterol-lowering medication commonly referred to as statin therapy.
Period: Overall Study
Arm/Group | Atorvastatin 40 mg Daily | Placebo Control
Started | 10 | 14
Completed | 10 | 13
Not Completed | 0 | 1
Not completed — Patient started prohibited medication | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Atorvastatin 40 mg Daily: Atorvastatin 40 mg daily x 16 weeks
- Placebo: Placebo daily x 16 weeks
- Total: Total of all reporting groups
Arm/Group | Atorvastatin 40 mg Daily | Placebo | Total
Number analyzed (Participants) | 10 | 14 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.0 (13.9) | 55.7 (5.3) | 53.3 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 1 | 4 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-hispanic | 8 | 13 | 21
  African-American | 1 | 1 | 2
  Asian | 1 | 0 | 1
History of hyperlipidemia [Number; unit: participants] | 4 | 2 | 6
History of hypertension [Count of Participants; unit: Participants] | 1 | 7 | 8
Obesity [Count of Participants; unit: Participants] | 2 | 6 | 8
Family history of early cardiovascular disease [Count of Participants; unit: Participants] | 1 | 1 | 2
mean modified Rodnan skin score [Mean (Standard Deviation); unit: points] — The modified Rodnan skin score (mRSS) measures skin thickness in 17 body areas. Each area is scored from 0 (no thickness) to 3 (bound down), and then summed. The mRSS range is 0-51. 0 is normal, and indicative of no skin thickening. Higher scores indicate greater skin thickening.
  points | 18.9 (9.6) | 22.8 (8.9) | 21.3 (9.2)
Mean EndoPAT reactive hyperemia index (RHI) [Mean (Standard Deviation); unit: units] — RHI ≤ 1.67 is abnormal and indicates endothelial dysfunction. A score of 1.67 or above suggests normal endothelial function. Results are presented as mean RHI +/- standard deviation.
  units | 1.36 (0.36) | 1.85 (1.20) | 1.46 (0.96)
Raynaud condition score (median, IQR) [Median (Inter-Quartile Range); unit: units on a scale] — The RCS is a self-assessment of Raynaud phenomenon activity using a 0-10 ordinal scale. Patients are asked to "please rate the difficulty you had today with your Raynaud condition by circling the appropriate number below". 0 indicates no difficulty, and 10 the most difficulty.
  units on a scale | 5.0 [3.0 to 7.5] | 2.0 [1.0 to 4.0] | 2.5 [1.0 to 4.5]
Raynaud symptom severity assessed by visual analog scale [Median (Inter-Quartile Range); unit: units on a scale] — This is a visual analog scale that is measured from 0-15 cm. 0 corresponds to no activity/severity, and 15 to the highest level.
  units on a scale | 4.0 [2.0 to 7.5] | 1.5 [0.5 to 3.0] | 2.3 [1.0 to 5.5]
Brachial % flow mediated dilation (%FMD) [Median (Inter-Quartile Range); unit: %] | 11.3 [7.4 to 14.7] | 10.3 [7.1 to 13.2] | 10.3 [7.3 to 13.6]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Improving Their EndoPAT Reactive Hyperemia Index (RHI) at the End-of-study (16 Weeks)
Description: EndoPAT is a proprietary device that assesses digital (microvascular) endothelial function during reactive hyperemia. A probe is placed on both index fingers. After 5 minutes of baseline observation, one arm is occluded for 5 minutes, while the other is not and serves as control. Output is the reactive hyperemia index (RHI), calculated as the post-to-pre occlusion signal ratio in the occluded side, "normalized to the control side and further corrected for baseline vascular tone" per Itamar Medical. There are no units. RHI ≤ 1.67 is abnormal and indicates endothelial dysfunction.
Time Frame: Change in RHI from baseline to 16 weeks expressed as the percentage of patients who improve (respond).
Population: The patient who did not complete the study had his data analyzed using last observation carried forward. Improvement was defined as an increase in the RHI from baseline to 16 weeks. Non-responders were defined as no change or worsening (decrease) in the RHI at 16 weeks. Results are expressed as a percentage
Measure: Count of Participants; unit: Participants
Arm/Group | Active Drug | Placebo Control
Number analyzed (Participants) | 10 | 14
Participants | 6 | 4

2. Secondary Outcome: Change in the Raynaud Condition Score (RCS) at 16 Weeks (End-of-study) From Baseline
Description: The Raynaud Condition Score is a patient-reported outcome of a single question regarding Raynaud severity. It is a visual analog scale with a results range of 0-100. A score of 0 us is no symptoms, and 100 severe symptoms. It is recommended by OMERACT for assessment of Raynaud phenomenon.
Time Frame: change in RCS from baseline to week 16
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Drug | Placebo Control
Number analyzed (Participants) | 10 | 14
score on a scale | -2.0 [-2.0 to 0] | 0 [-1.0 to 1.0]

3. Secondary Outcome: The Median Change in the Raynaud Phenomenon Visual Analog Scale (RP-VAS) Score at 16 Weeks (End-of-study) Compared to Baseline in the Atorvastatin and Placebo Groups.
Description: The RP-VAS scale measure ranges from 0-100, with 0 being no symptoms and 100 severe symptoms. Reported is the median and interquartile range of change between baseline and week 16 (end-of-study).
Time Frame: baseline to 16 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Drug | Placebo Control
Number analyzed (Participants) | 10 | 14
score on a scale | 0.5 [-1.5 to 6.0] | 0.0 [-1.0 to 1.5]

4. Secondary Outcome: % of Patients Who Improved Their Brachial Flow-mediation Dilation (%FMD) at 16 Weeks
Description: %FMD = change in brachial artery flow-mediation dilation between pre and post-ischemia. Baseline (pre-ischemia) is the reference to which percentage change is calculated.
  Result is expressed as the % of patients who had an improvement in their %FMD at 16 weeks compared to baseline.
Time Frame: baseline to 16 weeks
Population: For the patient with a SAE, data was treated as last observation carried forward
Measure: Count of Participants; unit: Participants
Arm/Group | Atorvastatin 40 mg Daily | Placebo
Number analyzed (Participants) | 10 | 14
Participants | 5 | 5

ADVERSE EVENTS:
Time Frame: 16 weeks plus 30 days after the end of intervention
Arm/Group | Atorvastatin 40 mg Daily | Placebo Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/10 | 1/14
Other Adverse Events (participants affected / at risk) | 0/10 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Atorvastatin 40 mg Daily (N=10) | Placebo Control (N=14)
Esophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Patient was diagnosed shortly before the end of the intervention period with esophageal cancer and pulmonary hypertension requiring vasodilators, which were prohibited in the protocol. The patient was withdrawn from the study.

LIMITATIONS AND CAVEATS:
This was a single-centered trial, and underpowered, as only 24 were enrolled with an initial goal of 30.

The groups were unbalanced for both the primary and secondary endpoint at baseline despite randomization.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT02370784/Prot_SAP_000.pdf